CLINICAL TRIAL: NCT04706312
Title: The Safety and Efficacy Assessment of Human Amniotic Mesenchymal Stem Cells(hAMSCs) Transplantation in Woman With Diminished Ovarian Reserve (DOR)
Brief Title: Transplantation of hAMSCs for Woman With DOR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SCR-03
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Diminished Ovarian Response
Keywords: Diminished ovarian response, human Amniotic Mesenchymal Stem Cells, Cell therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hAMSCs injection (Experimental): hAMSCs were injected via venous in the dorsum of hand.
  Interventions: Other: stem cells

INTERVENTIONS:
Other: stem cells — hAMSCs injection via venous in the dorsum of hand

SUMMARY:
Patients with Diminished ovarian response (DOR）have a poor in vitro fertilization（IVF） outcome, and is considered one of most challenging tasks in artificial reproductive treatment (ART). Stem cell therapies are rapidly progressing fields and have shown promise in treatment of lots of disease, including aging and premature ovarian failure. The purpose of this study is to determine the safety and efficacy of intra vein injection of human Amniotic Mesenchymal Stem Cells(hAMSCs) in women suffered from infertility caused by DOR.

DETAILED DESCRIPTION:
Patients with Diminished ovarian response (DOR）have a poor in vitro fertilization（IVF） outcome, and is considered one of most challenging tasks in artificial reproductive treatment (ART). Stem cell therapies are rapidly progressing fields and have shown immense promise in the treatment of lots of disease, including aging and premature ovarian failure. The purpose of this study is to determine the safety and efficacy of intra vein injection of human amniotic mesenchymal stem cells(hAMSCs) in women suffered from infertility caused by DOR. The hAMSCs were isolated and cultured in vitro and qualified by National Institutes for Food and Drug Control, China. The serum of each patient was kept and sent for laboratory test before the transplantation. The biomarkers of hAMSCs were detected again before transplantation. The hAMSCs were transplanted via venous in the dorsum of hand. The outcomes of patients were examined during and after the injection. The patients are monitored for hormones, follicles stimulated with minimal stimulation, number of oocyte retrieval and embryos In Vitro Fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

1. Women between35 and 45 years, who is diagnosed with Diminished Ovarian Reserve by Bologna criteria, (AFC≤7，or serum AMH level < 1.10ng/ml), and failed pregnancies in at least two cycles of In Vitro Fertilization(IVF) or Intracytoplasmic Sperm Injection(ICSI).
2. Willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Patients diagnosed with hereditary, immunological and iatrogenic premature ovarian failure
2. Patients allergy to blood products
3. Patients diagnosed with abnormal coagulation function
4. Patients diagnosed with uterine malformation
5. Patients undergoing Preimplantation Genetic Testing
6. Patients diagnosed with hydrosalpinx
7. Patients diagnosed with infectious diseases
8. Contraindications for In Vitro Fertilization-Embryo Transfer(IVF-ET) or pregnancy
9. Prior personal history of stem cell clinical trail or other clinical trails
10. Unwilling to comply with study protocol
11. Patients identified with high risk for stem cell injection

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability after hAMSCs injection. | Up to 12 months after first hAMSCs injection
  Safety and tolerability assessed by Adverse Events and serious during injection and adverse events (SAEs) after injection assessed by long term follow-up .
The ratio of transplantable embryo in DOR patients after hAMSCs injection. | Up to 12 months after first hAMSCs injection
  The ratio of transplantable embryo to normal fertilized embryos in DOR patients after hAMSCs injection.

SECONDARY OUTCOMES:
Ovarian function in DOR patients after hAMSCs injection. | Up to 12 months after first hAMSCs injection
  Anti-müllerian Hormone (AMH) serum level, Follicle Stimulating Hormone (FSH) serum level, Estradiol (E2) serum level, Luteinizing Hormone (LH)serum level on menstrual day 2/3 will be evaluated after injection. The number of antral follicles will be recorded by transvaginal ultrasound scan.
Outcomes of IVF in DOR patients after hAMSCs injection. | Up to 12 months after first hAMSCs injection
  The number of oocyte retrieval, fertilization rate , blastocyst formation rate, implantation rate, incidence of clinical pregnancy rate, after hAMSCs injection.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayin Liu, Doctor, Study Chair — First Affiliated Hospital, Nanjing Medical University
Locations (1):
- Clinical Center of Reproductive Medicine at the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No